CLINICAL TRIAL: NCT00089141
Title: A Randomized Study to Evaluate The Efficacy of Mycophenolate Mofetil Added to The Systemic Immunosuppressive Regimen First Used For Treatment of Chronic Graft-Versus-Host Disease
Brief Title: Mycophenolate Mofetil (MMF) for Treatment of Chronic Graft-versus-host Disease (GVHD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low probability of positive outcome
Sponsor: Martin, Paul (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Martin, Paul, Member, Fred Hutchinson Cancer Center
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1697.00; FHCRC-1697.00; ROCHE-FHCRC-1697.00; UMN-2004UC007; CDR0000378054 (Registry Identifier: PDQ)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2009-08-26 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2009-08

CONDITIONS: Cancer
Keywords: graft versus host disease; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; atypical chronic myeloid leukemia; blastic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic idiopathic myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; juvenile myelomonocytic leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated childhood rhabdomyosarcoma; previously treated myelodysplastic syndromes; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Graft vs Host Disease; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Multiple Myeloma; Carcinoma, Ovarian Epithelial; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Testicular Neoplasms; Breast Neoplasms | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate mofetil (Active Comparator): Patients receive oral mycophenolate mofetil twice daily.
  Interventions: Drug: mycophenolate mofetil
- Placebo (Placebo Comparator): Patients receive oral placebo twice daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: mycophenolate mofetil — Given orally
  Other Names: CellCept
  Arms: Mycophenolate mofetil
Drug: placebo — Given orally
  Other Names: Control
  Arms: Placebo

SUMMARY:
RATIONALE: Mycophenolate mofetil added to immunosuppressive treatment regimens may be effective in treating newly diagnosed chronic graft-versus-host disease caused by stem cell transplantation. It is not yet known whether immunosuppressive treatment regimens are more effective with or without mycophenolate mofetil in treating chronic graft-versus-host disease.

PURPOSE: This randomized phase III trial is studying whether the addition of mycophenolate mofetil improves the efficacy of immunosuppressive treatment regimens in patients with newly diagnosed chronic graft-versus-host disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of immunosuppressive treatment regimens with vs without mycophenolate mofetil in patients with newly diagnosed chronic graft-vs-host disease.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, prospective, multicenter study. Patients are stratified according to organ involvement of chronic graft-versus-host disease (GVHD) (single organ vs multiple organs) and transplant center. Patients are randomized to 1 of 2 treatment arms.

All patients receive usual therapy for chronic GVHD comprising oral prednisone twice daily and oral cyclosporine, oral tacrolimus or oral sirolimus twice daily until 2 weeks after the first evidence of improvement of symptoms of chronic GVHD.

* Arm I: Patients receive oral mycophenolate mofetil twice daily.
* Arm II: Patients receive oral placebo twice daily. In both arms administration of the study drug continues for 3 months after completion of prednisone and cyclosporine, tacrolimus or sirolimus in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then every 3 months.

Patients are followed every 3 months for 3-5 years.

PROJECTED ACCRUAL: A total of 230 patients (115 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed chronic-graft-versus host disease (GVHD)
* Systemic immunosuppressive treatment indicated AND no contraindication to treatment with mycophenolate mofetil
* Has undergone prior transplantation with any type of donor, hematopoietic stem cell graft, or conditioning regimen
* No clinical, laboratory, or image-based evidence known to be present at the time of enrollment and indicating a high probability of subsequent recurrent or progressive disease

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Not specified

Renal

* Not specified

Pulmonary

* No known bronchiolitis obliterans as a manifestation of chronic GVHD

Immunologic

* No fungal infection without radiographic evidence of improvement during continued antifungal therapy
* No cytomegalovirus (CMV) pneumonia without major radiographic evidence of improvement
* No other CMV infection without reduction of antigenemia or viral load during continued antiviral therapy
* No active disseminated varicella zoster viral infection
* No known hypersensitivity or allergy to MMF

Gastrointestinal

* Able to tolerate oral medication
* No lactose-intolerant children who are too young to swallow capsules
* No frank blood from the rectum
* No melena
* No known gastrointestinal ulceration

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Female patients must use 2 forms of contraception 4 weeks prior to, during, and for 6 weeks after completion of study treatment
* Not hospitalized at time of enrollment
* No rare, hereditary deficiency of hypoxanthine-guanine phosphoribosyl-transferase (HGPRT)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* Not specified

Endocrine therapy

* Prior treatment with prednisone or equivalent allowed provided the dose was ≤ 1.0 mg/kg/day at the time of enrollment
* Concurrent systemic glucocorticoids allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Prior mycophenolate mofetil (MMF) for prevention or treatment of acute GVHD allowed provided MMF was discontinued at least 2 weeks before the diagnosis of chronic GVHD was made
* No prior systemic treatment for chronic GVHD
* No prior treatment for chronic GVHD
* Concurrent antacids allowed provided there is at least a 2-hour interval before and after administration of MMF
* No other concurrent systemic immunosuppressive treatment except cyclosporine, tacrolimus or sirolimus

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2004-05; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Martin, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (16):
- United States (15):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Stanford Cancer Center, Stanford, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington
- Princess Margaret Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Martin PJ, Storer BE, Rowley SD, Flowers ME, Lee SJ, Carpenter PA, Wingard JR, Shaughnessy PJ, DeVetten MP, Jagasia M, Fay JW, van Besien K, Gupta V, Kitko C, Johnston LJ, Maziarz RT, Arora M, Jacobson PA, Weisdorf D. Evaluation of mycophenolate mofetil for initial treatment of chronic graft-versus-host disease. Blood. 2009 May 21;113(21):5074-82. doi: 10.1182/blood-2009-02-202937. Epub 2009 Mar 6. PMID 19270260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinic patients were recruited from May 2004 through June 2008.
Groups:
- Mycophenolate Mofetil: Patients receive oral mycophenolate mofetil 1000 mg twice daily.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil | Placebo
Started | 74 | 77
Completed | 56 | 53
Not Completed | 18 | 24
Not completed — Termination of trial | 18 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil | Placebo | Total
Number analyzed (Participants) | 74 | 77 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 68 | 71 | 139
  >=65 years | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.3) | 47.9 (13.3) | 48.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 41 | 40 | 81
Region of Enrollment [Number; unit: participants]
  United States | 73 | 75 | 148
  Canada | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Cure of Chronic GVHD Without Resorting to Secondary Systemic Therapy
Description: Withdrawal of all systemic immunosuppressive treatment after resolution of chronic GVHD, before death or onset of recurrent malignancy
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 11 | 10
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .22, Regression, Cox — P values are 2 sided and are based on likelihood ratio statistics; Analysis for all endpoints was stratified by number of affected organs and type of conditioning regimen; Hazard Ratio (HR) = 1.66, 95% CI [0.7 to 3.7] — For all analyses, MMF arm in numerator, and placebo arm in denominator. Hazard ratio estimate includes 3 efficacy success events that occurred after two years in the placebo arm

2. Secondary Outcome: Definitive Absence of Efficacy Success
Description: Administration of secondary systemic therapy for chronic GVHD, death during primary therapy, or onset of recurrent malignancy or bronchiolitis obliterans during primary therapy
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 45 | 40
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .03, Regression, Cox; Statistical analysis did not count treatment continuing beyond 2 years as efficacy failure (n = 2 in each arm); Hazard Ratio (HR) = 1.65, 95% CI [1.1 to 2.6]

3. Secondary Outcome: Open Label Systemic Treatment Because of Inadequate Response to Primary Therapy
Description: Administration of any systemic therapy other than the immunosuppressive agents used for initial treatment, because of persistent or progressive chronic graft-versus-host disease
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 24 | 25
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .55, Regression, Cox; Hazard Ratio (HR) = 1.19, 95% CI [0.7 to 2.1]

4. Secondary Outcome: Bronchiolitis Obliterans
Description: Development of bronchiolitis obliterans during treatment
Time Frame: within 4 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 5 | 4
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .48, Regression, Cox; Hazard Ratio (HR) = 1.61, 95% CI [0.4 to 6.0]

5. Secondary Outcome: Recurrent Malignancy
Description: Development of recurrent malignancy after enrollment in the study
Time Frame: within 4 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 17 | 10
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .17, Regression, Cox; adjusted for risk category; Hazard Ratio (HR) = 1.74, 95% CI [0.8 to 3.9]

6. Secondary Outcome: Non-relapse Mortality
Description: Death without prior development of recurrent malignancy
Time Frame: within 4 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 8 | 5
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .41, Regression, Cox; Hazard Ratio (HR) = 1.62, 95% CI [0.5 to 5.0]

7. Secondary Outcome: Death or Recurrent Malignancy
Description: Death due to any cause or development of recurrent malignancy at any time after enrollment
Time Frame: within 4 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 25 | 15
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .14, Regression, Cox; Hazard Ratio (HR) = 1.69, 95% CI [0.9 to 3.2]

8. Secondary Outcome: Death
Description: Death from any cause after enrollment in the study
Time Frame: within 4 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 19 | 10
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .10, Regression, Cox; Hazard Ratio (HR) = 1.99, 95% CI [0.9 to 4.3]

9. Secondary Outcome: Withdrawal of Prednisone
Description: Withdrawal of treatment with prednisone after improvement or resolution of chronic GVHD
Time Frame: within 4 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 30 | 33
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .34, Regression, Cox; Hazard Ratio (HR) = 1.28, 95% CI [.08 to 2.1]

10. Secondary Outcome: End of Systemic Treatment
Description: Withdrawal of all immunosuppressive treatment without recurrent malignancy
Time Frame: within 4 years
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Placebo
Number analyzed (Participants) | 74 | 77
participants | 15 | 15
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Placebo; Test type: Superiority or Other; p = .28, Regression, Cox; Hazard Ratio (HR) = 1.51, 95% CI [0.7 to 3.2]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No